CLINICAL TRIAL: NCT02877810
Title: Evidence-Based Tele-Emergency Network Grant Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: 678668; G01RH27872 (Other Grant/Funding Number: HRSA)
Record Dates: First submitted 2016-08-03; First posted 2016-08-24 (Estimated); Last update posted 2019-10-30 (Actual); Status verified 2019-10

CONDITIONS: Critical Illness
MeSH Terms: conditions — Critical Illness | interventions — Telemedicine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Telemedicine (Experimental): A consultation will be given for the care of a critically ill pediatric patient to a remote hospital emergency department physician by telemedicine, a live, interactive, audiovisual teleconferencing system, from a pediatric critical care physician.
  Interventions: Other: Telemedicine
- Telephone (Active Comparator): A consultation will be given for the care of a critically ill pediatric patient to a remote hospital emergency department physician by telephone, from a pediatric critical care physician..
  Interventions: Other: Telephone

INTERVENTIONS:
Other: Telemedicine — Telemedicine is a live, interactive, audiovisual teleconferencing system.
  Arms: Telemedicine
Other: Telephone — Consultations will be given over telephone.
  Arms: Telephone

SUMMARY:
The purpose of this study is to determine the impact of an existing tele-emergency care network on quality of care, appropriateness of care utilization, patient safety (medication errors), and cost effectiveness compared to telephone consultations from a healthcare system prospective.

DETAILED DESCRIPTION:
The investigators will use a novel cluster randomized unbalanced crossover trial design. When a new site is enrolled, the first approximately 6 months of the project will be a "ramp-up" period during which the protocol will be re-reviewed during a site visit to the participating EDs and random block assignments will be generated and delivered. The last 6 months will be reserved for data analysis, study closeout, and manuscript preparation. An intervening 2-year period will be divided into 4 six-month calendar time periods for carrying out the protocol and data collection. For each 6-month period, each ED will have a randomized treatment assignment for pediatric emergency and critical care consultations ("M" for telemedicine and "P" for telephone.) Participating EDs (the unit of randomization) will be stratified into two strata by size of ED and geographical location. EDs will then be randomized within-strata to one of the four unbalanced (3:1) crossover treatment assignment sequences, each consisting of a 6-month period: PMMM, MPMM, MMPM, or MMMP. During these assigned periods, the type of consultation being assigned will be strongly encouraged, but deviating from protocol (i.e., using telephone consultation when randomized to telemedicine, or the vice-versa) will be allowed as needed by the physicians. Data will be collected and abstracted through retrospective chart review.

ELIGIBILITY:
Inclusion Criteria:

* Children younger than or equal to 14 years of age at the time of their ED visit.

Exclusion Criteria:

* Children evaluated at the ED for non-medical reasons such as elective surgeries and social reasons (i.e., cases of possible endangerment) and other non-medical reasons.
* Children evaluated at the ED preoperatively, for elective surgical procedures.
* Children transferred to the ED from another hospital ED.
* Children transiently "held" in the ED in the process of a direct admission to the ward.

Max Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 696 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2018-08 (Actual); Study Completion 2019-08 (Actual)

PRIMARY OUTCOMES:
Quality of Care Implicit Review Instrument | Year 3
  The investigators hypothesize that children receiving care in EDs during periods of telemedicine use will receive higher quality of care than similar children who receive care during periods of telephone use. A previously validated 5-item implicit review instrument that measures 4 aspects of process of care in the ED, along with a fifth item assessing the overall quality of care provided to the patient will be used. The sum of the 5 item-specific scores will be aggregated from each reviewer to obtain a summary quality score for each medical record.
Pediatric Risk of Admission (PRISA II) | Year 3
  The investigators hypothesize that children receiving care in EDs during randomized periods of telemedicine use will be admitted more appropriately than similar children who receive care during periods randomized to telephone use. To compare the cohort of seriously ill children treated during the telephone and telemedicine time blocks, observed to expected (O/E) ratios will be calculated using an intention-to-treat framework.
Pediatric Emergency Assessment Tool (Re-PEAT) | Year 3
  The investigators hypothesize that children receiving care in EDs during randomized periods of telemedicine use will be transferred more appropriately than similar children who receive care during periods randomized to telephone use. The investigators will compare O/E ratios.
Medication Error Rate Instrument | Year 3
  The investigators hypothesize that children receiving care in EDs during periods of telemedicine use will experience fewer physician-related medication errors than similar children who receive care during periods of telephone use. A previously published instrument developed specifically to evaluate medication errors among children receiving care in the ED will be used.
Economic Efficiency Cost-Analysis | Year 3
  The investigators hypothesized that care provided to children in EDs during randomized periods of telemedicine use will be economically more efficient than care provided during randomized periods of telephone. Cost analysis will estimate return-on-investment indicating the cost saving amount per $1 investment in telemedicine compared to care without telemedicine.

CONTACTS AND LOCATIONS:
Overall Officials: James P Marcin, MD, MPH, Principal Investigator — University of California, Davis
Locations (1):
- University of California, Davis, Medical Center, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Marcin JP, Lieng MK, Mouzoon J, Sauers-Ford HS, Tancredi D, Cabri A, Pandya VA, Park AS, Kuppermann N. Telemedicine vs Telephone Consultations and Medication Prescribing Errors Among Referring Physicians: A Cluster Randomized Crossover Trial. JAMA Netw Open. 2024 Feb 5;7(2):e240275. doi: 10.1001/jamanetworkopen.2024.0275. PMID 38421649
- [Derived] Marcin JP, Sauers-Ford HS, Mouzoon JL, Haynes SC, Dayal P, Sigal I, Tancredi D, Lieng MK, Kuppermann N. Impact of Tele-Emergency Consultations on Pediatric Interfacility Transfers: A Cluster-Randomized Crossover Trial. JAMA Netw Open. 2023 Feb 1;6(2):e2255770. doi: 10.1001/jamanetworkopen.2022.55770. PMID 36780158